CLINICAL TRIAL: NCT04067609
Title: Postoperative Dexamethasone on Post-Cesarean Pain in Patients Using Medication Assisted Treatment (MAT)
Brief Title: Postoperative Dexamethasone on Post-Cesarean Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000025968; 000 (Other: CTGTY)
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post-Cesarean Pain; Cesarean Section Complications
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: a pilot double blind, placebo controlled randomized control trial using 40 subjects
Who Masked: Participant
Masking Description: double blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- patients receiving dexamethasone (Experimental): subjects will receive a single administration of either 0.1 mg/kg of intravenous dexamethasone in 90mL of normal saline
  Interventions: Drug: Dexamethasone
- placebo (Placebo Comparator): 100mL of normal saline (placebo) immediately upon the subjects' arrival to the Post Anesthesia Care Unit (PACU) after leaving the operating room from their scheduled c-section
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Dexamethasone — subjects will receive a single administration of either 0.1 mg/kg of intravenous dexamethasone in 90mL of normal saline
  Arms: patients receiving dexamethasone
Other: placebo — 100mL of normal saline (placebo)
  Arms: placebo

SUMMARY:
Investigating if giving post-operative dexamethasone to patients with a history of opioid use disorder on medication assisted treatment during pregnancy improves their pain scores and decreases their opioid use after cesarean section.

DETAILED DESCRIPTION:
For this study, the researchers are most interested in an option that would be able to be administered consistently (same time/same way): that labor nurses could give and without requiring the patient to have had an epidural placement. Further, Gabapentin, clonidine and ketamine are associated with CNS effects like sedation or confusion that could make health care providers less likely to be comfortable giving these women additional oxycodone due to possible worsened sedation or respiratory depression. Lastly, the researchers wanted to give a drug that both obstetricians and pediatricians were comfortable with from extensive use in our maternal population. Thus, a single administration IV dexamethasone was chosen for this study. Dexamethasone has been used as an adjunct for post-operative pain management in many types of surgeries. Although no large randomized trials exist, several small trials suggest an analgesic and opioid sparing effect of dexamethasone post-operatively for both pregnant and non-pregnanat patients; however these studies excluded patients on MAT

ELIGIBILITY:
Inclusion Criteria:

* English-speaking,
* History of opioid use disorder with current use of MAT during pregnancy,
* Scheduled for cesarean delivery for their current pregnancy for any indication [examples of elective c-section (decision made for c-section to be performed prior to onset of labor): fetal malpresentation, suspected macrosomia, prior c-section, abnormal placentation, patient preference],
* Negative toxicology screen upon admission to the hospital for their cesarean section, no prior administration of betamethasone for fetal lung maturity within 24h of their scheduled cesarean delivery

Exclusion Criteria:

* non-english speaking,
* screen positive for illicit substance(s) on their admission toxicology screen,
* require general anesthesia for their cesarean section due to maternal/fetal indication for non-anticipated urgency (thus no longer 'elective') or failure of adequate intra- operative pain control with spinal anesthesia,
* medical history including known cardiovascular disease, heart failure, uncontrolled hypertension, uncontrolled gestational diabetes or uncontrolled pregestational diabetes, active GI bleed or untreated peptic ulcer,
* untreated infectious diseases including tuberculosis, systemic candida

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women undergoing Cesarean section
Enrollment: 24 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Wesevich, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Receiving Dexamethasone | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Receiving Dexamethasone | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (4.1) | 31.7 (3.6) | 31.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Gravidity [Mean (Standard Deviation); unit: pregnancies] | 3.8 (1.1) | 3.8 (1.5) | 3.8 (1.3)
Living Children [Mean (Standard Deviation); unit: children] | 1.3 (0.6) | 1.6 (1.1) | 1.4 (0.9)
Body Mass Index (BMI) at Delivery [Mean (Standard Deviation); unit: kg/m^2] | 35.9 (8.3) | 30.2 (5.2) | 33.1 (7.3)
Number of Prior Cesarean Sections [Mean (Standard Deviation); unit: Cesarean Sections] | 1 (0.9) | 1.3 (1) | 1.1 (0.9)
Insurance Type [Count of Participants; unit: Participants]
  Medicaid | 12 | 11 | 23
  Private | 0 | 1 | 1
Medication Type [Count of Participants; unit: Participants]
  Methadone | 9 | 10 | 19
  Subutex | 3 | 2 | 5
Breastfeeding [Count of Participants; unit: Participants]
  Yes | 11 | 8 | 19
  No | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score
Description: Pain scores via the standardly used and accepted Visual Analog Scale ranging from 1 (lowest) to 10 (highest).
Time Frame: 24, 48, 72 and 96 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Receiving Dexamethasone | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  0-24 hours post-op | 4.1 (2.9) | 4.2 (3.2)
  25-48 hours post-op | 5.1 (2.3) | 5.2 (2.0)
  49-72 hours post-op | 4.6 (2.2) | 4.5 (1.9)
  73-96 hours post-op | 3.9 (2.4) | 3.8 (2.0)

2. Secondary Outcome: Change of Morphine Use
Description: Comparison of total morphine dose equivalents used by the patient during this period will be examined. The total morphine dose equivalents will be calculated from the total narcotic dose and appropriate conversion (i.e. dilaudid dose to morphine dose equivalents). This will be calculated as a total daily dose for the hospital stay and an average dose/d over the entire hospital stay. These 2 separate calculations will be used because it is presumed that narcotic use will decrease with each day post-op. Calculating an average dose/d over the entire hospital stay will account for women who are discharged on different postoperative days.
Time Frame: 24, 48 and 72 hours post-op
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents/day
Arm/Group | Patients Receiving Dexamethasone | Placebo
Number analyzed (Participants) | 12 | 12
Morphine milligram equivalents/day
  0-24 hours post-op | 32.3 (30.6) | 34.4 (28.9)
  25-48 hours post-op | 38.3 (29.6) | 44.5 (34.2)
  49-72 hours post-op | 14.3 (22.9) | 20.6 (32)

ADVERSE EVENTS:
Time Frame: up to 96 hours post-op
Arm/Group | Patients Receiving Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT04067609/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT04067609/ICF_001.pdf